CLINICAL TRIAL: NCT04237792
Title: A PHASE 3/4 RANDOMIZED, DOUBLE-BLIND, DOSE-RANGING STUDY OF THE SAFETY AND EFFICACY OF DEXMEDETOMIDINE (DEX) USED WITH PROPOFOL (PRO) AS NEEDED FOR PROCEDURAL SEDATION OF PEDIATRIC SUBJECTS ≥1 MONTH TO <17 YEARS OF AGE UNDERGOING MRI SCANS
Brief Title: Safety and Efficacy of Dexmedetomidine (DEX) for Sedation of Subjects ≥1 Month to <17 Years Undergoing MRI Scans
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: C0801039
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: MRI Sedation
Keywords: procedural sedation; dexmedetomidine; propofol; MRI
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- dexmedetomidine low dose group (Experimental): low dose of dexmedetomidine to be given
  Interventions: Drug: dexmedetomidine; Drug: propofol
- dexmedetomidine middle dose group (Experimental): middle dose of dexmedetomidine to be given
  Interventions: Drug: dexmedetomidine; Drug: propofol
- dexmedetomidine high dose group (Experimental): high dose of dexmedetomidine to be given
  Interventions: Drug: dexmedetomidine; Drug: propofol

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine low, middle and high doses are provided as an intravenous bolus loading dose followed by an intravenous maintenance dose infusion throughout the MRI scan
Drug: propofol — propofol IV administration will be given if needed to maintain sedation

SUMMARY:
This is a randomized, double-blind, dose-ranging study of the efficacy and safety of dexmedetomidine (DEX) when used with propofol as needed, for procedural sedation of pediatric subjects ≥1 month to <17 years of age undergoing MRI scans in the US and Japan.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subject ≥1 month and <17 years of age.
2. American Society of Anesthesiologists (ASA) Physical Status I, II or III.
3. Requires non-intubated, spontaneous breathing, moderate to deep sedation (NI MDS) for a magnetic resonance imaging (MRI) study with an intensivist, anesthesiologist or other proceduralist in attendance.
4. Duration of the MRI scan is expected to take at least 20 minutes but no more than 3 hours to complete

Key Exclusion Criteria:

1. Pregnant female subjects (including those with an indeterminate or positive pregnancy test); breastfeeding female subjects.
2. Weight on Day 1 before randomization is less than the 10th percentile of weight for age and sex in the US and Japan or is greater than the 95th percentile of weight for age and sex in the US or greater than the 97th percentile of weight for age and sex in Japan based on sponsor-provided growth charts.
3. Planned medical procedure during the MRI scan or post-MRI recovery period.
4. Requires endotracheal intubation or laryngeal mask airway (LMA).
5. Known allergy to eggs, egg products, soybeans or soybean products.
6. SpO2 <93 % on room air -

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (16):
  - Arkansas Children's, Little Rock, Arkansas
  - Lucile Packard Children's Hospital, Stanford, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - Baptist Health - Wolfson Children's Hospital, Jacksonville, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta-Egleston, Atlanta, Georgia
  - IU Health Riley Hospital for Children, Indianapolis, Indiana
  - University of Michigan, C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - M Health Fairview University of Minnesota Medical Center - West Bank, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - University Hospitals Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - The Children's Hospital at OUMC, Oklahoma City, Oklahoma
  - Children's Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Japan (7):
  - Ibaraki Children Hospital, Mito, Ibaraki
  - Shikoku Medical Center for Children and Adults, Zentsujichó, Kagawa-ken
  - Osaka Women's and Children's Hospital, Izumi-shi, Osaka
  - Shizuoka Children's Hospital, Shizuoka, Shizuoka
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Osaka City General Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0801039

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total 141 participants were screened. Out of 141 participants, only 128 participants who met eligibility criteria signed the informed consent document, were enrolled and randomized. Out of 128 randomized participants, 6 participants were not treated.
Pre-assignment Details: Pediatric participants were administered with dexmedetomidine (DEX), and with propofol (PRO) as needed, for procedural sedation for magnetic resonance imaging (MRI) scans.
Groups:
- Low Dose: Age >=1 Month to <2 Years: Day 1: Participants aged >=1 month to <2 years, were randomized to receive a loading dose of DEX 0.5 microgram per kilogram (mcg/kg) over 10 minutes as intravenous (IV) infusion followed by continuous maintenance dose of DEX 0.5 mcg/kg/hour IV. If an adequate level of sedation was not achieved, participants were co-administered with PRO IV per physical investigator (PI) clinical judgment. MRI scan started on achieving an adequate sedation level. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours. Treatment PRO first bolus strength would be 500 mcg/kg and then maintenance infusion at 50 mcg/kg/min. Participants were monitored for a minimum of 1 hour after completion of MRI scan. Day 2: Participants were followed up after 24 hours (+/- 2 hours) post discontinuation of DEX. Participants had a long-term follow-up contact via phone call at 28 to 31 days post last administration of study drug.
- Middle Dose: Age >=1 Month to <2 Years: Day 1: Participants aged >=1 month to <2 years, were randomized to receive a loading dose of DEX 1 mcg/kg over 10 minutes as IV infusion followed by continuous maintenance dose of DEX 1 mcg/kg/hour IV. If an adequate level of sedation was not achieved, participants were co-administered with PRO IV per PI clinical judgment. MRI scan started on achieving an adequate sedation level. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours. Treatment PRO first bolus strength would be 500 mcg/kg and then maintenance infusion at 50 mcg/kg/min. Participants were monitored for a minimum of 1 hour after completion of MRI scan. Day 2: Participants were followed up after 24 hours (+/- 2 hours) post discontinuation of DEX. Participants had a long-term follow-up contact via phone call at 28 to 31 days post last administration of study drug.
- High Dose: Age >=1 Month to <2 Years: Day 1: Participants aged >=1 month to <2 years, were randomized to receive a loading dose of DEX 1.5 mcg/kg over 10 minutes as IV infusion followed by continuous maintenance dose of DEX 1.5 mcg/kg/hour IV. If an adequate level of sedation was not achieved, participants were co-administered with PRO IV per PI clinical judgment. MRI scan started on achieving an adequate sedation level. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours. Treatment PRO first bolus strength would be 500 mcg/kg and then maintenance infusion at 50 mcg/kg/min. Participants were monitored for a minimum of 1 hour after completion of MRI scan. Day 2: Participants were followed up after 24 hours (+/- 2 hours) post discontinuation of DEX. Participants had a long-term follow-up contact via phone call at 28 to 31 days post last administration of study drug.
- Low Dose: Age >=2 Years to <17 Years: Day 1: Participants aged >=2 years to <17 years, were randomized to receive a loading dose of DEX 0.5 mcg/kg over 10 minutes as IV infusion followed by continuous maintenance dose of DEX 0.5 mcg/kg/hour IV. If an adequate level of sedation was not achieved, participants were co-administered with PRO IV per PI clinical judgment. MRI scan started on achieving an adequate sedation level. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours. Treatment PRO first bolus strength would be 500 mcg/kg and then maintenance infusion at 50 mcg/kg/min. Participants were monitored for a minimum of 1 hour after completion of MRI scan. Day 2: Participants were followed up after 24 hours (+/- 2 hours) post discontinuation of DEX. Participants had a long-term follow-up contact via phone call at 28 to 31 days post last administration of study drug.
- Middle Dose: Age >=2 Years to <17 Years: Day 1: Participants aged >=2 years to <17 years, were randomized to receive a loading dose of DEX 1.2 mcg/kg over 10 minutes as IV infusion followed by continuous maintenance dose of DEX 1 mcg/kg/hour IV. If an adequate level of sedation was not achieved, participants were co-administered with PRO IV per PI clinical judgment. MRI scan started on achieving an adequate sedation level. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours. Treatment PRO first bolus strength would be 500 mcg/kg and then maintenance infusion at 50 mcg/kg/min. Participants were monitored for a minimum of 1 hour after completion of MRI scan. Day 2: Participants were followed up after 24 hours (+/- 2 hours) post discontinuation of DEX. Participants had a long-term follow-up contact via phone call at 28 to 31 days post last administration of study drug.
- High Dose: Age >=2 Years to <17 Years: Day 1: Participants aged >=2 years to <17 years, were randomized to receive a loading dose of DEX 2 mcg/kg over 10 minutes as IV infusion followed by continuous maintenance dose of DEX 1.5 mcg/kg/hour IV. If an adequate level of sedation was not achieved, participants were co-administered with PRO IV per PI clinical judgment. MRI scan started on achieving an adequate sedation level. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours. Treatment PRO first bolus strength would be 500 mcg/kg and then maintenance infusion at 50 mcg/kg/min. Participants were monitored for a minimum of 1 hour after completion of MRI scan. Day 2: Participants were followed up after 24 hours (+/- 2 hours) post discontinuation of DEX. Participants had a long-term follow-up contact via phone call at 28 to 31 days post last administration of study drug.
Period: Treatment (Day 1)
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years
Started | 21 | 22 | 20 | 23 | 21 | 21
Treated With DEX | 20 | 21 | 18 | 22 | 21 | 20
Completed | 19 | 21 | 17 | 22 | 20 | 18
Not Completed | 2 | 1 | 3 | 1 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Not treated | 1 | 1 | 2 | 1 | 0 | 1
Period: MRI Scan (Day 1)
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years
Started | 20 (DEX infusion could be discontinued during MRI scan, if clinically indicated.) | 21 | 18 (DEX infusion could be discontinued during MRI scan, if clinically indicated.) | 22 | 21 (DEX infusion could be discontinued during MRI scan, if clinically indicated.) | 20 (DEX infusion could be discontinued during MRI scan, if clinically indicated.)
Completed | 20 | 21 | 18 | 22 | 21 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Post MRI Scan Recovery (Day 1)
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years
Started | 20 | 21 | 18 | 22 | 21 | 20
Completed | 20 | 21 | 18 | 22 | 21 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up (FU) (Day 2)
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years
Started | 20 | 21 | 18 | 22 | 21 | 20
Completed | 20 | 21 | 18 | 22 | 21 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Long Term FU (Any Day From Day 29 to 32)
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years
Started | 20 | 21 | 18 | 22 | 21 | 20
Completed | 20 | 21 | 18 | 22 | 21 | 20
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who received any amount of DEX.
Groups:
- Low Dose: Age >=1 Month to <2 Years: Day 1: Participants aged >=1 month to <2 years, were randomized to receive a loading dose of DEX 0.5 mcg/kg over 10 minutes as IV infusion followed by continuous maintenance dose of DEX 0.5 mcg/kg/hour IV. If an adequate level of sedation was not achieved, participants were co-administered with PRO IV per PI clinical judgment. MRI scan started on achieving an adequate sedation level. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours. Treatment PRO first bolus strength would be 500 mcg/kg and then maintenance infusion at 50 mcg/kg/min. Participants were monitored for a minimum of 1 hour after completion of MRI scan. Day 2: Participants were followed up after 24 hours (+/- 2 hours) post discontinuation of DEX. Participants had a long-term follow-up contact via phone call at 28 to 31 days post last administration of study drug.
- Total: Total of all reporting groups
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Total
Number analyzed (Participants) | 20 | 21 | 18 | 22 | 21 | 20 | 122
Age, Continuous [Mean (Standard Deviation); unit: Years] | 0.99 (0.612) | 0.90 (0.488) | 0.96 (0.384) | 6.68 (2.922) | 7.40 (3.230) | 6.63 (3.277) | 4.02 (3.743)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 8 | 11 | 10 | 9 | 59
  Male | 8 | 12 | 10 | 11 | 11 | 11 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 7 | 0 | 3 | 3 | 19
  Not Hispanic or Latino | 15 | 18 | 11 | 22 | 17 | 17 | 100
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Asian | 3 | 8 | 4 | 11 | 8 | 7 | 41
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 1 | 1 | 0 | 2 | 2 | 8
  White | 10 | 8 | 11 | 10 | 9 | 9 | 57
  More than one race | 1 | 0 | 0 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 3 | 2 | 2 | 0 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants at the DEX High Dose Versus Low Dose in the Combined Age Cohorts Who Did Not Require Concomitant PRO to Complete MRI
Description: Percentage of participants who did not require PRO to complete MRI scan in the combined age cohorts are reported in this outcome measure.
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: FAS included all randomized participants who received any amount of DEX.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- High Dose: Combined Age: Participants aged >=1 month to <2 years and >=2 years to <17 years were randomized to receive a loading dose of DEX 1.5 mcg/kg over 10 minutes followed by maintenance dose of DEX 1.5 mcg/kg/hour and a loading dose of DEX 2 mcg/kg over 10 minutes followed by maintenance dose of DEX 1.5 mcg/kg/hour respectively. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
- Low Dose: Combined Age: Participants aged >=1 month to <2 years and >=2 years to <17 years were randomized to receive a loading dose of DEX 0.5 mcg/kg over 10 minutes followed by maintenance dose of DEX 0.5 mcg/kg/hour respectively. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
Arm/Group | High Dose: Combined Age | Low Dose: Combined Age
Number analyzed (Participants) | 38 | 42
Percentage of participants | 63.2 [46.0 to 78.0] | 14.3 [5.0 to 29.0]
Statistical Analysis 1: Comparison: High Dose: Combined Age vs Low Dose: Combined Age; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.03 to 0.29]

2. Secondary Outcome: Percentage of Participants at the DEX High Dose Versus Low Dose in Each Age Cohort Who Did Not Require Concomitant PRO to Complete MRI
Description: Percentage of participants who did not require PRO to complete MRI scan in each age cohort are reported in this outcome measure.
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: FAS included all randomized participants who received any amount of DEX.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- High Dose: Age >=1 Month to <2 Years: Participants aged >=1 month to < 2 years, were randomized to receive a loading dose of DEX 1.5 mcg/kg over 10 minutes followed by maintenance dose of DEX 1.5 mcg/kg/hour. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
- Low Dose: Age >=1 Month to <2 Years: Participants aged >=1 month to < 2 years, were randomized to receive a loading dose of DEX 0.5 mcg/kg over 10 minutes followed by maintenance dose of DEX 0.5 mcg/kg/hour. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
- High Dose: Age >=2 Years to <17 Years: Participants aged >=2 years to <17 years, were randomized to receive a loading dose of DEX 2 mcg/kg over 10 minutes followed by maintenance dose of DEX 1.5 mcg/kg/hour. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
- Low Dose: Age >=2 Years to <17 Years: Participants aged >=2 years to <17 years, were randomized to receive a loading dose of DEX 0.5 mcg/kg over 10 minutes followed by maintenance dose of DEX 0.5 mcg/kg/hour. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
Arm/Group | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=1 Month to <2 Years | High Dose: Age >=2 Years to <17 Years | Low Dose: Age >=2 Years to <17 Years
Number analyzed (Participants) | 18 | 20 | 20 | 22
Percentage of participants | 50.0 [26.0 to 74.0] | 15.0 [3.0 to 38.0] | 75.0 [51.0 to 91.0] | 13.6 [3.0 to 35.0]
Statistical Analysis 1: Comparison: High Dose: Age >=1 Month to <2 Years vs Low Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.022, Mantel Haenszel; Odds Ratio (OR) = 0.18, 95% CI 2-sided [0.04 to 0.82]
Statistical Analysis 2: Comparison: High Dose: Age >=2 Years to <17 Years vs Low Dose: Age >=2 Years to <17 Years; Test type: Other; p < 0.001, Mantel Haenszel; Odds Ratio (OR) = 0.05, 95% CI 2-sided [0.01 to 0.26]

3. Secondary Outcome: Percentage of Participants at the DEX Middle Dose vs Low Dose and High Dose vs Middle Dose in Each Age Cohort and Combined Age Cohorts Who Did Not Require Concomitant PRO to Complete MRI
Description: Percentage of participants who did not require PRO to complete MRI scan in each age cohort and combined age cohorts are reported in this outcome measure.
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: FAS included all randomized participants who received any amount of DEX.
Measure: Number; unit: Percentage of participants
Groups:
- Middle Dose: Age >=1 Month to <2 Years: Participants aged >=1 month to < 2 years, were randomized to receive a loading dose of DEX 1 mcg/kg over 10 minutes followed by maintenance dose of DEX 1 mcg/kg/hour. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
- Middle Dose: Age >=2 Years to <17 Years: Participants aged >=2 years to <17 years, were randomized to receive a loading dose of DEX 1.2 mcg/kg over 10 minutes followed by maintenance dose of DEX 1 mcg/kg/hour. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
- Middle Dose: Combined Age: Participants aged >=1 month to <2 years and >=2 years to <17 years were randomized to receive a loading dose of DEX 1 mcg/kg over 10 minutes followed by maintenance dose of DEX 1 mcg/kg/hour and a loading dose of DEX 1.2 mcg/kg over 10 minutes followed by maintenance dose of DEX 1 mcg/kg/hour respectively. If adequate sedation was not achieved PRO was co-administered. DEX and PRO (if needed) continued till completion of MRI scan. MRI scan was expected to complete in not more than 3 hours.
Arm/Group | High Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | Low Dose: Age >=1 Month to <2 Years | High Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | Low Dose: Age >=2 Years to <17 Years | High Dose: Combined Age | Middle Dose: Combined Age | Low Dose: Combined Age
Number analyzed (Participants) | 18 | 21 | 20 | 20 | 21 | 22 | 38 | 42 | 42
Percentage of participants | 50.0 | 9.5 | 15.0 | 75.0 | 61.9 | 13.6 | 63.2 | 35.7 | 14.3
Statistical Analysis 1: Comparison: High Dose: Age >=1 Month to <2 Years vs Middle Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.006, Mantel Haenszel; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.02 to 0.59]
Statistical Analysis 2: Comparison: Middle Dose: Age >=1 Month to <2 Years vs Low Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.597, Mantel Haenszel; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.25 to 11.27]
Statistical Analysis 3: Comparison: High Dose: Age >=2 Years to <17 Years vs Middle Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.374, Mantel Haenszel; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.14 to 2.07]
Statistical Analysis 4: Comparison: Middle Dose: Age >=2 Years to <17 Years vs Low Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.001, Mantel Haenszel; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.02 to 0.44]
Statistical Analysis 5: Comparison: High Dose: Combined Age vs Middle Dose: Combined Age; Test type: Other; p = 0.015, Mantel Haenszel; Odds Ratio (OR) = 0.32, 95% CI 2-sided [0.13 to 0.81]
Statistical Analysis 6: Comparison: Middle Dose: Combined Age vs Low Dose: Combined Age; Test type: Other; p = 0.024, Mantel Haenszel; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.10 to 0.87]

4. Secondary Outcome: Percentage of Time at Target Pediatric Sedation State Scale (PSSS) Score of 2 After the Administration of the DEX Loading Dose and During the DEX Maintenance Infusion - By Age Cohort and Combined Age
Description: In this outcome measure percentage of time for which participant had maintained PSSS score of 2 was reported. PSSS score ranges from 0 to 5, where 0= sedation with abnormal physiologic parameters requiring acute intervention, 1= sedation with normal vital signs, but requiring airway intervention, 2= no movement during procedure, no frown, no verbalization of complaint indicating no pain and anxiety, 3= no movement during procedure but expression of pain and anxiety on face, verbalization of complaint, requiring help positioning, 4= movement during procedure requiring gentle immobilization for positioning, verbalization of some discomfort or stress, but no crying or shouting that expresses stress or objection, 5= movement impeding proceduralist and requiring forceful immobilization, crying or shouting during procedure, but vocalization not required. Higher score indicated less sedation.
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: FAS included all randomized participants who received any amount of DEX. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Low Dose: Combined Age | Middle Dose: Combined Age | High Dose: Combined Age
Number analyzed (Participants) | 20 | 21 | 18 | 22 | 20 | 20 | 42 | 41 | 38
Percentage of time | 77.5 (15.94) | 82.5 (12.04) | 87.8 (23.93) | 76.8 (18.36) | 92.2 (9.72) | 94.1 (12.22) | 77.2 (17.04) | 87.2 (11.88) | 91.1 (18.71)
Statistical Analysis 1: Comparison: Middle Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.021, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Low Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.007, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Low Dose: Age >=1 Month to <2 Years vs Middle Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.225, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Middle Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.213, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Low Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Low Dose: Age >=2 Years to <17 Years vs Middle Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Middle Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.011, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Low Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Low Dose: Combined Age vs Middle Dose: Combined Age; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Time From the Start of DEX Loading Dose Infusion to the Time of First PRO Bolus Infusion - By Age Cohort and Combined Age
Description: Participants who did not have PRO administered were censored.
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: FAS included all randomized participants who received any amount of DEX.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Low Dose: Combined Age | Middle Dose: Combined Age | High Dose: Combined Age
Number analyzed (Participants) | 20 | 21 | 18 | 22 | 21 | 20 | 42 | 42 | 38
Minutes | 16.0 [15.0 to 21.0] | 17.0 [16.0 to 25.0] | 62.0 [19.0 to NA] — Upper value of 95 % confidence interval (CI) could not be estimated due to less number of participants with event. | 16.5 [15.0 to 25.0] | NA [31.0 to NA] — Median and upper value of 95 % CI could not be estimated due to less number of participants with event. | NA [72.0 to NA] — Median and upper value of 95 % CI could not be estimated due to less number of participants with event. | 16.0 [15.0 to 20.0] | 31.5 [17.0 to 64.0] | NA [45.0 to NA] — Median and upper value of 95 % CI could not be estimated due to less number of participants with event.
Statistical Analysis 1: Comparison: Middle Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.016, Log Rank
Statistical Analysis 2: Comparison: Low Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.005, Log Rank
Statistical Analysis 3: Comparison: Low Dose: Age >=1 Month to <2 Years vs Middle Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.368, Log Rank
Statistical Analysis 4: Comparison: Middle Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.358, Log Rank
Statistical Analysis 5: Comparison: Low Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.000, Log Rank
Statistical Analysis 6: Comparison: Low Dose: Age >=2 Years to <17 Years vs Middle Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.001, Log Rank
Statistical Analysis 7: Comparison: Middle Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.020, Log Rank
Statistical Analysis 8: Comparison: Low Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.000, Log Rank
Statistical Analysis 9: Comparison: Low Dose: Combined Age vs Middle Dose: Combined Age; Test type: Other; p = 0.005, Log Rank

6. Secondary Outcome: Emergence Time - By Age Cohort and Combined Age
Description: Emergence time: time from the end of the MRI scan to when the participant met a Modified Aldrete score >=9. Participants who were withdrawn or discharged without reaching a Modified Aldrete score >=9, were censored, time computed from end of MRI scan to time of the last clinical assessment (vital signs). Zero minute was used as the censored time if no vital signs were taken during the post-MRI recovery period. Modified Aldrete score: validated observational medical scoring system that allowed verbal prompts for the measurement of recovery after anesthesia (post anesthesia) which included items: activity, respiration, circulation, consciousness, and oxygenation. Each item was scored from 0 to 2, higher scores signified better recovery. The scores of each item were summed to obtain a total score of 0 to 10, where higher scores indicated well recovered participant post anesthesia.
Time Frame: Post MRI scan on Day 1 up to 24 hours
Population: FAS included all randomized participants who received any amount of DEX.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Low Dose: Combined Age | Middle Dose: Combined Age | High Dose: Combined Age
Number analyzed (Participants) | 20 | 21 | 18 | 22 | 21 | 20 | 42 | 42 | 38
Minutes | 30.0 [6.0 to 59.0] | 41.0 [34.0 to 54.0] | 38.0 [12.0 to 51.0] | 35.0 [21.0 to 49.0] | 46.0 [25.0 to 64.0] | 50.0 [35.0 to 62.0] | 35.0 [21.0 to 41.0] | 42.5 [35.0 to 52.0] | 45.5 [35.0 to 54.0]
Statistical Analysis 1: Comparison: Middle Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.884, Log Rank
Statistical Analysis 2: Comparison: Low Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.662, Log Rank
Statistical Analysis 3: Comparison: Low Dose: Age >=1 Month to <2 Years vs Middle Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.236, Log Rank
Statistical Analysis 4: Comparison: Middle Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.733, Log Rank
Statistical Analysis 5: Comparison: Low Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.128, Log Rank
Statistical Analysis 6: Comparison: Low Dose: Age >=2 Years to <17 Years vs Middle Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.165, Log Rank
Statistical Analysis 7: Comparison: Middle Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.752, Log Rank
Statistical Analysis 8: Comparison: Low Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.139, Log Rank
Statistical Analysis 9: Comparison: Low Dose: Combined Age vs Middle Dose: Combined Age; Test type: Other; p = 0.051, Log Rank

7. Secondary Outcome: Number of Participants Who Received PRO - By Age Cohort and Combined Age
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: FAS included all randomized participants who received any amount of DEX.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Low Dose: Combined Age | Middle Dose: Combined Age | High Dose: Combined Age
Number analyzed (Participants) | 20 | 21 | 18 | 22 | 21 | 20 | 42 | 42 | 38
Participants | 17 | 19 | 9 | 19 | 8 | 5 | 36 | 27 | 14

8. Secondary Outcome: Total Amount (mcg Per kg) of Concomitant PRO Required to Successfully Complete MRI - By Age Cohort and Combined Age
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg per kg
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Low Dose: Combined Age | Middle Dose: Combined Age | High Dose: Combined Age
Number analyzed (Participants) | 17 | 19 | 9 | 19 | 8 | 5 | 36 | 27 | 14
mcg per kg | 4012.1 (2334.66) | 4730.3 (3398.21) | 2822.8 (1593.84) | 5559.2 (4038.95) | 5001.9 (4093.70) | 4513.0 (4620.56) | 4828.6 (3390.42) | 4810.7 (3538.71) | 3426.4 (2973.00)
Statistical Analysis 1: Comparison: Middle Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.124, ANOVA
Statistical Analysis 2: Comparison: Low Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.186, ANOVA
Statistical Analysis 3: Comparison: Low Dose: Age >=1 Month to <2 Years vs Middle Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.470, ANOVA
Statistical Analysis 4: Comparison: Middle Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.845, ANOVA
Statistical Analysis 5: Comparison: Low Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.621, ANOVA
Statistical Analysis 6: Comparison: Low Dose: Age >=2 Years to <17 Years vs Middle Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.747, ANOVA
Statistical Analysis 7: Comparison: Middle Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.218, ANOVA
Statistical Analysis 8: Comparison: Low Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.181, ANOVA
Statistical Analysis 9: Comparison: Low Dose: Combined Age vs Middle Dose: Combined Age; Test type: Other; p = 0.984, ANOVA

9. Secondary Outcome: Body Weight/Time Adjusted Total Amount (Per kg Per Minute) of Concomitant PRO Required to Successfully Complete MRI - By Age Cohort and Combined Age
Time Frame: Up to maximum of 3 hours during MRI scan on Day 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg per kg per minute
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Low Dose: Combined Age | Middle Dose: Combined Age | High Dose: Combined Age
Number analyzed (Participants) | 17 | 19 | 9 | 19 | 7 | 4 | 36 | 26 | 13
mcg per kg per minute | 59.43 (18.625) | 71.38 (32.895) | 47.41 (14.454) | 81.28 (38.406) | 74.70 (24.487) | 76.36 (47.656) | 70.96 (32.243) | 72.28 (30.418) | 56.31 (30.007)
Statistical Analysis 1: Comparison: Middle Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.048, ANOVA
Statistical Analysis 2: Comparison: Low Dose: Age >=1 Month to <2 Years vs High Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.106, ANOVA
Statistical Analysis 3: Comparison: Low Dose: Age >=1 Month to <2 Years vs Middle Dose: Age >=1 Month to <2 Years; Test type: Other; p = 0.196, ANOVA
Statistical Analysis 4: Comparison: Middle Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.940, ANOVA
Statistical Analysis 5: Comparison: Low Dose: Age >=2 Years to <17 Years vs High Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.824, ANOVA
Statistical Analysis 6: Comparison: Low Dose: Age >=2 Years to <17 Years vs Middle Dose: Age >=2 Years to <17 Years; Test type: Other; p = 0.678, ANOVA
Statistical Analysis 7: Comparison: Middle Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.129, ANOVA
Statistical Analysis 8: Comparison: Low Dose: Combined Age vs High Dose: Combined Age; Test type: Other; p = 0.160, ANOVA
Statistical Analysis 9: Comparison: Low Dose: Combined Age vs Middle Dose: Combined Age; Test type: Other; p = 0.872, ANOVA

ADVERSE EVENTS:
Time Frame: Day 1 up to maximum of 31 days after last dose of study drug (up to maximum of 32 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. The safety analysis set consisted of all randomized participants who received any amount of DEX. Safety data was presented by dose level, overall (combined two age cohorts) and within each age cohort.
Groups:
- Combined Dose: Age >=1 Month to <2 Years: Participants were randomized to receive a loading dose of DEX 0.5 mcg/kg (low dose), 1 mcg/kg (middle dose), and 1.5 mcg/kg (high dose) over 10 minutes followed by maintenance dose of DEX 0.5 mcg/kg/hour (low dose), 1 mcg/kg/hour (middle dose), and 1.5 mcg/kg/hour (high dose).
- Combined Dose: Age >=2 Years to <17 Years: Participants were randomized to receive a loading dose of DEX 0.5 mcg/kg (low dose), 1.2 mcg/kg (middle dose), and 2 mcg/kg (high dose) over 10 minutes followed by maintenance dose of DEX 0.5 mcg/kg/hour (low dose), 1 mcg/kg/hour (middle dose), and 1.5 mcg/kg/hour (high dose).
Arm/Group | Low Dose: Age >=1 Month to <2 Years | Middle Dose: Age >=1 Month to <2 Years | High Dose: Age >=1 Month to <2 Years | Combined Dose: Age >=1 Month to <2 Years | Low Dose: Age >=2 Years to <17 Years | Middle Dose: Age >=2 Years to <17 Years | High Dose: Age >=2 Years to <17 Years | Combined Dose: Age >=2 Years to <17 Years
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/18 | 0/59 | 0/22 | 0/21 | 0/20 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/18 | 0/59 | 0/22 | 0/21 | 1/20 | 1/63
Other Adverse Events (participants affected / at risk) | 19/20 | 20/21 | 17/18 | 56/59 | 19/22 | 19/21 | 19/20 | 57/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose: Age >=1 Month to <2 Years (N=20) | Middle Dose: Age >=1 Month to <2 Years (N=21) | High Dose: Age >=1 Month to <2 Years (N=18) | Combined Dose: Age >=1 Month to <2 Years (N=59) | Low Dose: Age >=2 Years to <17 Years (N=22) | Middle Dose: Age >=2 Years to <17 Years (N=21) | High Dose: Age >=2 Years to <17 Years (N=20) | Combined Dose: Age >=2 Years to <17 Years (N=63)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose: Age >=1 Month to <2 Years (N=20) | Middle Dose: Age >=1 Month to <2 Years (N=21) | High Dose: Age >=1 Month to <2 Years (N=18) | Combined Dose: Age >=1 Month to <2 Years (N=59) | Low Dose: Age >=2 Years to <17 Years (N=22) | Middle Dose: Age >=2 Years to <17 Years (N=21) | High Dose: Age >=2 Years to <17 Years (N=20) | Combined Dose: Age >=2 Years to <17 Years (N=63)
Bradycardia (Cardiac disorders) | 9 | 12 | 13 | 34 | 15 | 12 | 14 | 41
Rebound tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 3 | 1 | 0 | 1 | 2
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Syringomyelia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 16 | 12 | 47 | 14 | 11 | 10 | 35
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 6 | 3 | 0 | 1 | 4
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diastolic hypertension (Vascular disorders) | 1 | 3 | 3 | 7 | 2 | 0 | 1 | 3
Diastolic hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 9 | 12 | 9 | 30 | 2 | 5 | 8 | 15
Hypotension (Vascular disorders) | 9 | 6 | 3 | 18 | 4 | 5 | 3 | 12
Systolic hypertension (Vascular disorders) | 0 | 3 | 1 | 4 | 1 | 2 | 2 | 5
Withdrawal hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT04237792/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/92/NCT04237792/SAP_001.pdf